CLINICAL TRIAL: NCT05135156
Title: Lung Transplant Resources for Education and Decision-making for Your Cystic Fibrosis (READY): A Pilot Randomized Controlled Trial
Brief Title: Lung Transplant READY Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Kathleen Ramos, Assistant Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: STUDY00011578; 1R03HL158728-01 (NIH)
Record Dates: First submitted 2021-11-22; First posted 2021-11-26 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Lung Transplantation; Lung Disease; Decision Support Tool
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Access to an investigator-designed web-based educational resource with information about lung transplant for two weeks.
  Interventions: Behavioral: Investigator-designed lung transplant education resource (Research Intervention)
- Control (Active Comparator): Access to a publicly available web-based educational resource with information about transplant for two weeks.
  Interventions: Behavioral: Publicly available transplant education resource (Attention Control)

INTERVENTIONS:
Behavioral: Investigator-designed lung transplant education resource (Research Intervention) — Participants will access the investigator-designed educational resource via their login to a secure website. After two weeks, participants will gain access to the publicly available website (attention control) and will have an additional two weeks of access to both of these resources.
  Arms: Intervention
Behavioral: Publicly available transplant education resource (Attention Control) — Participants will access the publicly available education resource via their login to a secure website. After two weeks, participants will gain access to the investigator-designed educational resource (research intervention) and will have an additional two weeks of access to both of these resources.
  Arms: Control

SUMMARY:
Lung transplant is an option for treating end-stage lung disease in cystic fibrosis (CF). More than half of people with CF who die without a lung transplant were never referred for consideration. Patient preference not to undergo lung transplant may account for 25-40% of decisions to defer referral. Increasing awareness of lung transplant among people with CF, and promoting understanding of the risks and benefits of transplant, can potentially reduce the number of people with CF who die without a lung transplant.

The CF Foundation (CFF) lung transplant referral guidelines were developed to optimize the timing of referral for lung transplant. These guidelines recommend annual conversations with CF patients once their forced expiratory volume in one second (FEV1) is <50% predicted. Considering lung transplant as a treatment option ahead of when it is medically needed will allow more time to learn about lung transplant and address any barriers to lung transplant that may exist.

Investigators are interested in understanding how people with CF use lung transplant educational resources and how one prepares for having discussions and/or making decisions about lung transplant as a treatment option for advanced CF. The purpose of this study is to test whether a research website improves patient preparedness for discussions about lung transplant.

Study involvement will span 4 weeks and study procedures will involve the following:

* Three Zoom interview sessions (30-60 minutes each)
* Survey assessments
* Access to a research website that contains educational resources about lung transplant (goal of 4 hours of use over the 4 week study period)

DETAILED DESCRIPTION:
Lung transplant is an option for treating end-stage lung disease in cystic fibrosis (CF). In the United States, more CF patients with forced expiratory volume in 1 second (FEV1) less than 30% of predicted die each year than undergo lung transplant. More than half of people with CF who die without lung transplant were never referred for consideration, with patients of lower socioeconomic status disproportionately impacted by limited access to lung transplant. Patient preference not to undergo lung transplant may account for 25-40% of decisions to defer referral. The CF Foundation established lung transplant referral guidelines that recommend individuals with CF have annual conversations about lung transplant with their CF doctor once their FEV1 is less than 50% of predicted. Considering lung transplant as a treatment option ahead of when it is medically needed will allow more time to learn about lung transplant and address any barriers to lung transplant that may exist. By introducing an educational resource that can increase awareness of lung transplant among patients, and promote understanding of the risks and benefits of lung transplant, investigators aim to empower people with CF to take part in shared decision-making with their CF providers which could reduce the number of people with CF who die without lung transplant.

Based on prior research, investigators have developed a novel lung transplant decision support tool that addresses patient-identified knowledge gaps and provides personalized educational content to help people with CF prepare for lung transplant discussions and decisions. The decision support tool couples real-life CF patient experiences of lung transplant in the form of personal narratives with up-to-date, CF-specific, and guideline-based medical information about lung transplant.

The overall research objectives for this pilot study are to test the efficacy of the decision support tool to improve patient preparedness for shared decision making about lung transplant and knowledge about lung transplant, and to evaluate the impact on mental health outcomes (depression and anxiety). The new website will be compared against an attention control website (UNOS.org) to better understand how people with CF use and rank different educational resources' utility. The central hypothesis is that use of the new decision support tool that incorporates disease severity data (FEV1 % predicted, supplemental oxygen use, exacerbations) to identify relevant personal narratives and guideline-based educational content will increase a patient's preparedness to engage in discussions about lung transplant beyond the standard information presented on UNOS.org.

The pilot study will be a randomized controlled trial. Participants will be randomized 1:1 to one of two educational resources, described above, stratified by FEV1 category (FEV1 30-50% or FEV1 <30% of predicted). Baseline surveys will evaluate knowledge about lung transplant, a Likert scale rating of preparedness for lung transplant discussions, decisional conflict about lung transplant, and mental health. Baseline interviews will address perspectives on lung transplant as a treatment option for CF and the role of newer CF therapies in the decision making process about lung transplant. For two weeks, participants will have access to one of two educational resources via a login to a secure research website. At 2 weeks, there will be a study visit that includes repeated surveys from baseline and the Preparedness for Shared Decision Making (PrepDM) Scale, along with a second brief interview. After the 2-week study visit, participants will have access to both educational resources via individual login to the secure research website. At 4 weeks, there will be a study visit to repeat the surveys and interview. Throughout the 4 weeks, web analytics will be captured at the individual level to determine usage patterns for both educational resources.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis
* FEV1 less than or equal to 50% predicted (unless referred per MD recommendation)

Exclusion Criteria:

* Patients unable to provide informed consent
* Patients who are lung transplant recipients
* Unable to read or understand English to complete surveys or access the websites (currently only available in English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Ramos, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) may be shared with other researchers for secondary analyses with the approval of the appropriate Human Subjects Division(s) and the study's principal investigator (PI).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available after publication of the results of the primary analyses of the study. The data will be available for up to 3 years after the end of the study.
Access Criteria: Qualified researchers with appropriate clinical research training and/or mentorship will be allowed to have access to IPD after approval is obtained from Human Subjects Division(s) and the study PI.

REFERENCES:
- [Background] Ramos KJ, Smith PJ, McKone EF, Pilewski JM, Lucy A, Hempstead SE, Tallarico E, Faro A, Rosenbluth DB, Gray AL, Dunitz JM; CF Lung Transplant Referral Guidelines Committee. Lung transplant referral for individuals with cystic fibrosis: Cystic Fibrosis Foundation consensus guidelines. J Cyst Fibros. 2019 May;18(3):321-333. doi: 10.1016/j.jcf.2019.03.002. Epub 2019 Mar 27. PMID 30926322
- [Background] Leard LE, Holm AM, Valapour M, Glanville AR, Attawar S, Aversa M, Campos SV, Christon LM, Cypel M, Dellgren G, Hartwig MG, Kapnadak SG, Kolaitis NA, Kotloff RM, Patterson CM, Shlobin OA, Smith PJ, Sole A, Solomon M, Weill D, Wijsenbeek MS, Willemse BWM, Arcasoy SM, Ramos KJ. Consensus document for the selection of lung transplant candidates: An update from the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2021 Nov;40(11):1349-1379. doi: 10.1016/j.healun.2021.07.005. Epub 2021 Jul 24. PMID 34419372
- [Background] Ramos KJ, Hobler MR, Engelberg RA, Curtis JR, Zander MI, Howard SS, Goss CH, Aitken ML. Addressing lung transplant with adults with cystic fibrosis: A qualitative analysis of patients' perspectives and experiences. J Cyst Fibros. 2019 May;18(3):416-419. doi: 10.1016/j.jcf.2019.04.007. Epub 2019 Apr 17. PMID 31003953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A screening survey was advertised at 15 CF Centers in the United States who agreed to approach their adult CF patients with an FEV1 <50% predicted to share information about our study. Survey respondents could 'opt in' to being contacted about additional research opportunities related to lung transplant. We also approached CF patients at the University of Washington Adult CF Center who had an FEV1 <50% predicted. Recruitment occurred from December 2021 to November 2022.
Pre-assignment Details: A total of 52 participants consented. Of these, 2 were lost to follow up and 50 were randomized to study arms, 25 per arm.
Groups:
- Consented, Not Randomized: Participants who consented but were not randomized
Period: Overall Study
Arm/Group | Intervention | Control | Consented, Not Randomized
Started | 25 | 25 | 2
Completed | 25 | 25 | 0
Not Completed | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [30 to 40] | 40 [34 to 49] | 37 [31 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 10 | 16 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 23 | 25 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Community of Concern (Yes/No) [Count of Participants; unit: Participants] — Participants were considered to belong to a Community of Concern if they met one or more of the following criteria: Medicaid insurance, High school education or less, non-White race, Hispanic ethnicity.
  Participants | 18 | 13 | 31
Taking CFTR modulator [Count of Participants; unit: Participants] | 24 | 24 | 48
Current FEV1 %predicted [Count of Participants; unit: Participants]
  41-50% | 7 | 13 | 20
  30-40% | 14 | 8 | 22
  <30% | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Participants Completing 2-week Study Visit
Description: The co-primary endpoint is feasibility, which will be defined as successful if 90% of enrolled participants complete the 2-week study visit (regardless of study arm).
Time Frame: Measured at 2-week study visit
Measure: Count of Participants; unit: Participants
Groups:
- Consented, Not Randomized: Consented but lost to follow up prior to baseline study visit
Arm/Group | Intervention | Control | Consented, Not Randomized
Number analyzed (Participants) | 25 | 25 | 2
Participants | 25 | 25 | 0

2. Primary Outcome: Preparedness for Shared Decision Making (PrepDM) Scale
Description: The co-primary endpoint is an intention-to-treat assessment of the difference in mean Preparedness for Shared Decision Making (PrepDM) Scale in the intervention versus control arms of the study at the 2-week study visit. Scores range on a scale from 0 to 100 with higher scores indicating a higher perceived level of preparation for decision making.
Time Frame: Measured at 2-week study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
score on a scale | 71 (16) | 57 (23)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.02, Regression, Linear; Mean Difference (Final Values) = 14, 95% CI 2-sided [3 to 25] — Difference = intervention - control

3. Secondary Outcome: Confidence-weighted True False Knowledge About Lung Transplant (14-question Investigator-designed Survey)
Description: Difference in mean confidence-weighted true false (CTF) knowledge score will be measured in the intervention versus control arms of the study. CTF scoring adds points for certainty in correct responses and deducts points for certainty in incorrect responses. Participants receive +2 points when "sure" about a correct response, +1 if unsure about a correct response, -1 if unsure about an incorrect response and -2 if sure about an incorrect response. For a 14-item knowledge test, the maximum score is +28 and the minimum score is -28, with higher scores indicating more knowledge about lung transplant.
Time Frame: Measured at 2-week study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
score on a scale | 11.6 (6.0) | 8.8 (7.4)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.15, Regression, Linear; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-1.0 to 6.6] — Difference = intervention - control

4. Secondary Outcome: Decisional Conflict Scale
Description: Decisional Conflict Scale change will be measured from the baseline study visit to the 2-week study visit. The intention-to-treat analysis will compare mean change in the Decisional Conflict Scale between the intervention and control arms of the study. Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict].
Time Frame: Baseline to 2-week study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
score on a scale | -12 (17) | -11 (17)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.81, Regression, Linear; Mean Difference (Net) = -1.2, 95% CI 2-sided [-10.9 to 8.5] — Estimation parameter is regression parameter comparing intervention to control

5. Secondary Outcome: Likert-scale Rating of Preparedness to Discuss Lung Transplant (0-4)
Description: Likert rating of preparedness will be measured at the 2-week study visit (0=Don't know, 1= Not at all prepared, 2 = A little prepared, 3 = Moderately prepared, 4 = Very prepared). The intention-to-treat analysis will compare mean Likert-scale rating between the intervention and control arms of the study.
Time Frame: Measured at 2-week study visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
units on a scale | 3.4 (0.7) | 3.1 (0.9)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.15, Regression, Linear; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.1 to 0.8] — Difference = intervention - control

6. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: PHQ-9 is a scale that measures symptoms of depression in the prior 2 weeks on a 0-27 scale, with higher scores indicating worsening depression and a score of 10 or higher consistent with a diagnosis of depression. Investigators will assess the difference in mean PHQ-9 score in the intervention versus control arms of the study at the 2-week study visit.
Time Frame: Measured at 2-week study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
score on a scale | 5.6 (5.2) | 4.8 (4.8)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.54, Regression, Linear; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-2.0 to 3.7] — Estimation parameter is regression parameter comparing intervention to control

7. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: PHQ-9 is a scale that measures symptoms of depression in the prior 2 weeks on a 0-27 scale, with higher scores indicating worsening depression and a score of 10 or higher consistent with a diagnosis of depression. Investigators will determine the proportion with new PHQ-9 score greater than or equal to 10 in each arm.
Time Frame: Measured at 2-week study visit
Measure: Number; unit: proportion of participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
proportion of participants | 0.16 | 0.12

8. Secondary Outcome: Generalized Anxiety Disorder 7-item (GAD-7) Scale
Description: GAD-7 is a scale that measures symptoms of anxiety in the prior 2 weeks on a 0-21 scale, with higher scores indicating worsening anxiety and a score of 10 or higher consistent with a diagnosis of generalized anxiety disorder. Investigators will assess the difference in mean GAD-7 score in the intervention versus control arms of the study at the 2-week study visit.
Time Frame: Measured at 2-week study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
score on a scale | 4.6 (4.1) | 4.3 (4.3)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.82, Regression, Linear; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-2.1 to 2.7] — Difference = intervention - control

9. Secondary Outcome: Generalized Anxiety Disorder 7-item (GAD-7) Scale
Description: GAD-7 is a scale that measures symptoms of anxiety in the prior 2 weeks on a 0-21 scale, with higher scores indicating worsening anxiety and a score of 10 or higher consistent with a diagnosis of generalized anxiety disorder. Investigators will determine the proportion with new GAD-7 score greater than or equal to 10 in each arm.
Time Frame: Measured at 2-week study visit
Measure: Number; unit: proportion of participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
proportion of participants | 0.08 | 0.16

10. Other Pre Specified Outcome: 4-week Assessment of Preparedness for Shared Decision Making (PrepDM) Scale
Description: The PrepDM Scale will be measured for all participants with respect to the investigator-designed educational resource (research intervention) and mean score will be compared for participants in the intervention (4 weeks of exposure) versus control arms (2 weeks of exposure). PrepDM scores range on a scale from 0 to 100 with higher scores indicating a higher perceived level of preparation for decision making.
Time Frame: Measured at 4-week study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
score on a scale | 72 (22) | 77 (17)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.44, Regression, Linear; Mean Difference (Final Values) = -4, 95% CI 2-sided [-15 to 7] — Estimation parameter is regression parameter comparing intervention to control

11. Other Pre Specified Outcome: 4-week Assessment for Confidence-weighted True False Knowledge About Lung Transplant (14-question Investigator-designed Survey)
Description: Change in confidence-weighted true false knowledge about lung transplant (14-question investigator-designed survey with minimum possible score -28 and maximum possible score 28; higher scores indicate more knowledge about lung transplant) will be assessed from immediately prior to intervention exposure to the end of exposure time. For participants in the intervention arm, this represents change from baseline to 4-weeks. For participants in the Attention Control arm, this represents change from 2-week to 4-week study visits. The statistical analysis will compare mean change in the knowledge score from baseline to 4 weeks between study arms. This compares the effect of 4-week exposure to Take on Transplant [intervention arm] vs. 2-week exposure [control arm] on improvement in knowledge scores.
Time Frame: Measured at Baseline, 2-week study visit, 4-week study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
score on a scale | 4.4 (4.2) | 1.2 (4.2)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.31, Regression, Linear; Mean Difference (Net) = 1.3, 95% CI 2-sided [-1.3 to 3.9] — Estimation parameter is regression parameter comparing intervention to control

12. Other Pre Specified Outcome: 4-week Assessment for Decisional Conflict Scale
Description: Change in Decisional Conflict Scale (scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict]) will be assessed from immediately prior to intervention exposure to the end of exposure time. For participants in the intervention arm, this represents change from baseline to 4-weeks. For participants in the Attention Control arm, this represents change from 2-week to 4-week study visits. The statistical analysis will compare mean change in Decisional Conflict Scale from baseline to 4 weeks between study arms. This compares the effect of 4-week exposure to Take on Transplant [intervention arm] vs. 2-week exposure [control arm] on improvement in knowledge scores.
Time Frame: Measured at Baseline, 2-week study visit, 4-week study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
score on a scale | -16.4 (16.4) | -10.4 (21.4)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.42, Regression, Linear; Mean Difference (Net) = 5.0, 95% CI 2-sided [-7.4 to 17.4] — Difference = intervention - control; Estimation parameter is regression parameter comparing intervention to control

13. Other Pre Specified Outcome: 4-week Assessment for Likert-scale Rating of Preparedness to Discuss Lung Transplant
Description: Evaluate the proportion "Very prepared" at baseline, 2 weeks and 4 weeks in the intervention and control arms. Compare proportions across study arms at each time point.
Time Frame: Measured at baseline, 2-week and 4-week study visits
Measure: Number; unit: proportion of participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
proportion of participants
  Baseline | 0.52 | 0.40
  2 weeks | 0.52 | 0.40
  4 weeks | 0.76 | 0.60
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — Pearson's chi-squared test of independence; p = 0.39, Chi-squared — p=0.39 at baseline, 0.39 at 2 weeks and 0.23 at 4 weeks

14. Other Pre Specified Outcome: Time Spent Using the Research Website
Description: Median time spent using the research website from baseline to 2 weeks will be compared across study arms. Further, time spent using the investigator-designed website will be assessed as a predictor of: 1. change in confidence-weighted true false knowledge about lung transplant (14-question investigator-designed survey) from baseline to 2-week study visit, 2. change in Likert preparedness from baseline to 2-week study visit, 3. change in Decisional Conflict Scale from baseline to 2-week study visit, and 4. mean PrepDM Scale at 2-weeks.
Time Frame: Baseline to 2-week study visit
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 25
minutes | 133 [88 to 179] | 142 [81 to 215]
Statistical Analysis 1: Comparison: Intervention; Outcome = change in confidence-weighted true false knowledge about lung transplant (14-question investigator-designed survey) from baseline to 2-week study visit; Test type: Superiority; p = 0.91, Regression, Linear; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.84 to 0.94] — Parameters are for a 60-minute greater amount of time spent on the website (range was 21-418 minutes in the first 2 weeks)
Statistical Analysis 2: Comparison: Intervention; Outcome = change in Likert preparedness to discuss transplant from baseline to 2-week study visit; Test type: Superiority; p = 0.53, Regression, Linear; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.08 to 0.16] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Intervention; Outcome = change in Decisional Conflict Scale from baseline to 2-week study visit; Test type: Superiority; p = 0.04, Regression, Linear; Mean Difference (Net) = -4.3, 95% CI 2-sided [-8.4 to -0.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: Intervention; Test type: Superiority; p = 0.74, Regression, Linear — Outcome = mean PrepDM Scale at 2-weeks; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-3.6 to 5.0] — [estimate comment as in outcome 14, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during Zoom study visits (baseline, 2 weeks, 4 weeks).
Groups:
- Intervention: Investigator-designed lung transplant education resource (Research Intervention)
- Control: Publicly available transplant education resource (Attention Control)
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 2/25 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=25) | Control (N=25)
Possible suicidality endorsed on PHQ-9 (Psychiatric disorders) | 2 (3) | 1 (1) — For the purposes of this study, participant report of possible suicidality on the PHQ-9 (positive response to question #9) is an immediately reportable AE, even if it is not an SAE. PHQ-9 is only administered during Zoom study visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT05135156/Prot_SAP_ICF_000.pdf